CLINICAL TRIAL: NCT02626598
Title: A Study Evaluating Blended Belotero for the Treatment of Etched-in Fine Facial Lines
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Skin Care and Laser Physicians of Beverly Hills (Other)
Collaborators: Merz Aesthetics Inc. (Industry)
Responsible Party: Principal Investigator, Derek H. Jones, M.D., MD, Skin Care and Laser Physicians of Beverly Hills
Other Study IDs: IIS2202
Record Dates: First submitted 2015-11-30; First posted 2015-12-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Rhytidosis Facialis
Keywords: facial wrinkles; photoaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treated patients: Patients treated with blended Belotero for etched-in fine lines of the cutaneous lip, and/or radial cheek area, and/or nasolabial folds, and/or melolabial folds, and/or forehead area will be evaluated with photographs, physician ratings, and patient improvement assessments.
  Interventions: Device: Blended Belotero

INTERVENTIONS:
Device: Blended Belotero — Belotero blended with 0.1 cc of 1% lidocaine with epinephrine per 1.0 cc Belotero will be injected to etched in fine facial lines
  Other Names: Treated patients

SUMMARY:
This is a single center study for adult females or males ages 25 to 75 years who are seeking treatment for etched-in fine lines of the cutaneous lip, and/or radial cheek area, and/or nasolabial folds, and/or melolabial folds, and/or forehead. The purpose of this study is to evaluate blended Belotero for the treatment of etched-in fine facial lines and to monitor for adverse events.

DETAILED DESCRIPTION:
This is a study to evaluate the effects of Belotero blended with 0.1 cc of 1% lidocaine with epinephrine per 1.0 cc of Belotero in the treatment of etched-in fine facial lines. 30 adults scheduled to have blended Belotero injected into fine lines of the cutaneous lip, and/or radial cheek area, and/or nasolabial folds, and/or melolabial folds, and/or forehead will be evaluated. The blended Belotero will be injected intradermally into these etched-in fine lines. The patients will be given diary cards to document potential adverse events. 2 weeks after receiving injections of the blended Belotero the subjects will return to have photographs taken, have their treated fine lines evaluated, and complete a self assessment questionnaire. Touch-up injections are common clinical practice and if additional touch-ups would improve their result, those subjects can be re-treated at this visit. Those subjects who are touched up will return to the clinic for an additional follow up visit and photographs 2 weeks later. All subjects will return to the clinic 12 weeks and 24 weeks after their last injection for photographs and evaluations. Improvement assessments will be made by investigator ratings at each visit. Investigator ratings for the cutaneous lip and the forehead area are based on the Merz Aesthetic Validated Assessment Scales. Investigator ratings for the radial cheek area, nasolabial folds, and melolabial folds are based on the Validated Lemperle Facial Wrinkle Scales.

ELIGIBILITY:
Inclusion Criteria:

* Adult females and males, aged 25-75 years.
* Subjects must be seeking treatment for etched-in fine lines of the cutaneous lip area, and/or radial cheek area, and/or nasolabial fold area, and/or melolabial fold area, and/or forehead area.
* Subjects must have one or more etched-in fine line on the cutaneous lip area, and/or radial cheek area, and/or nasolabial fold area, and/or melolabial fold area, and/or forehead area.
* Subjects must have been deemed eligible by the treating physician and be scheduled for treatment of etched-in fine facial lines with Belotero blended with lidocaine with epinephrine.
* Subjects must be willing to defer any other cosmetic procedures in the treatment area while in the study. They can continue using topicals with retinoids, retinol, beta hydroxy acids, or alpha hydroxyl acids if they were previously using these topicals for at least 3 months prior to starting the study, but they should not initiate cosmetic treatments with new topicals during the study period. They should not have cosmetic treatments such as chemical peels, microdermabrasion, microneedling procedures, laser procedures, botulinum toxin injections, or other injectable filler therapy in the treatment area during the study period.
* Subjects must be willing and able to provide written informed consent in English
* Subjects must be willing and able to follow the procedures outlined in this protocol.

Exclusion Criteria:

* Subjects who are pregnant.
* Subjects with previous permanent injectable filler therapy to the treatment area.
* Subjects with previous non-permanent injectable filler therapy to the treatment area within the past year.
* Subjects with previous botulinum toxin injections in the treatment area within the past 6 months.
* Subjects with severe baseline facial lines in the treatment area with a score of 5 based on the Validated Lemperle Facial Wrinkle Scales.
* Subjects with visible scars in the treatment area that may affect evaluation of response and/or quality of photography in the opinion of the investigator.
* Known allergy or sensitivity to any of the treatment injections or their components, including or known or suspected lidocaine hypersensitivity.
* Subjects with an infection in the treatment area.
* Subjects are not to undergo any additional cosmetic procedures in the treatment area during the study period.
* Subjects with a history of poor cooperation, non-compliance with medical treatment, or unrealiability.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a single-center observational study of adult females and males ages 25 to 75 years who are scheduled to have treatment with Belotero blended with lidocaine with epinephrine, as is common in clinical practice for etched-in fine lines of the cutaneous lip, and/or radial cheek area, and/or nasolabial folds, and/or melolabial folds, and/or forehead area. After reviewing the risks and benefits of the procedure, the patient will sign a clinical consent form prior to treatment. If the patient is amenable to participate in the study and agrees to have pre and post treatment photographs and evaluations completed, they will proceed to sign the research consent form and will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Investigator Fine Facial Line Evaluations (Merz Aesthetic Validated Assessment Scales for cutaneous lip and the forehead and Validated Lemperle Facial Wrinkle Scales for the radial cheek, nasolabial folds, and melolabial folds) | 24-26 weeks
  Investigator evaluations and ratings of fine facial lines will be made at each visit. Investigator ratings for the cutaneous lip and the forehead area are based on the Merz Aesthetic Validated Assessment Scales. Investigator ratings for the radial cheek area, nasolabial folds, and melolabial folds are based on the Validated Lemperle Facial Wrinkle Scales.

SECONDARY OUTCOMES:
Patient Diary Cards Documenting Adverse Events | 2-4 weeks
  Patients will be given diary cards to document any potential adverse events for 2 weeks after each treatment.
Subject Improvement Evaluations of Treated Facial Lines | 24-26 weeks
  Subject improvement evaluations will be made at each visit with exception to the first visit. Subjects will rate the percent improvement of the treated facial lines (0-25% Improvement, 25-49% Improvement, 50-74% Improvement, or 75-100% Improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Derek H Jones, MD, Principal Investigator — Skin Care and Laser Physicians of Beverly Hills
Locations (1):
- Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California, United States

REFERENCES:
- [Background] Carruthers A, Carruthers J, Hardas B, Kaur M, Goertelmeyer R, Jones D, Rzany B, Cohen J, Kerscher M, Flynn TC, Maas C, Sattler G, Gebauer A, Pooth R, McClure K, Simone-Korbel U, Buchner L. A validated grading scale for forehead lines. Dermatol Surg. 2008 Nov;34 Suppl 2:S155-60. doi: 10.1111/j.1524-4725.2008.34364.x. PMID 19021673
- [Background] Lemperle G, Holmes RE, Cohen SR, Lemperle SM. A classification of facial wrinkles. Plast Reconstr Surg. 2001 Nov;108(6):1735-50; discussion 1751-2. doi: 10.1097/00006534-200111000-00048. PMID 11711957
- [Background] Moradi A, Shirazi A, Moradi-Poehler J, Turner J, Howell DJ. A blinded, randomized, split-face pilot study of bruising and pain with hyaluronic acid for correction of perioral lines using no lidocaine, lidocaine alone, and lidocaine and epinephrine. Aesthet Surg J. 2015 May;35(4):443-55. doi: 10.1093/asj/sjv043. PMID 25908703
- [Background] Narins RS, Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, de Maio M, Mohrmann C, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Breitscheidel L, Carruthers A. Validated assessment scales for the lower face. Dermatol Surg. 2012 Feb;38(2 Spec No.):333-42. doi: 10.1111/j.1524-4725.2011.02247.x. PMID 22316189